CLINICAL TRIAL: NCT01210794
Title: The Influence of Different Food Componente on Zinc Absorption in Young Adults Consuming Zinc Fortified Porridges Prepared From Maize, Beans and Sorghum: a Series of Six Similar Randomized, Single-blind Studies
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: ETH Zurich, Human Nutrition Laboratory (Unknown)
Responsible Party: Sponsor
Other Study IDs: HNL/CTC08-09
Record Dates: First submitted 2010-09-27; First posted 2010-09-28 (Estimated); Last update posted 2012-01-10 (Estimated); Status verified 2012-01

CONDITIONS: Study Not Related to a Disease. Nutrition Study Without Drug Administration.

INTERVENTIONS:
Procedure:  — The influence of different food components on zinc absorption in young adults consuming zinc fortified porridges prepared from maize, beans and sorghum

SUMMARY:
The influence of different food componente on zinc absorption in young adults consuming zinc fortified porridge's prepared from maize, beans and sorghum: a series of six similar randomized, single-blind studies.

ELIGIBILITY:
Inclusion criteria:

1. Male or female of 18 to 45 years old
2. Body Mass Index in the range of 19 to 25
3. No mineral and vitamin supplements two weeks prior to the study and during the whole duration of the study

Exclusion criteria:

1. Any metabolic, gastrointestinal or chronic disease (according to the subjects own statement)
2. Long-term medication during the whole study (except for contraceptives)
3. Smoking
4. Pregnancy
5. Lactating
6. Earlier participation in any other clinical study within the last 30 days

   * Subject Withdrawal:

     * Incomplete consumption of test meal
     * Missing of test meal Missing of iv dose
     * Incomplete urine collection (studies 2-6); exceptions to be discussed for study 1
     * No blood sample at start of study
     * Consumption of food within 3 hours after iv dose - to be evaluated
     * Vomiting within 3 hours after test meal administration - to be evaluated
     * Sick subjects and subjects taking any medication during study - to be evaluated (postponement of test meal possible)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Study not related to a disease. Nutrition study without drug drug administration. Investigation on the influence of different food components on zinc absorption in young adults consuming zinc fortified porridges prepared from maize, beans and sorghum.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2009-03; Study Completion 2010-06

CONTACTS AND LOCATIONS:
Overall Officials: Rita Wegmueller, Dr, Principal Investigator — ETH Zurich, Human Nutrition Laboratory
Locations (1):
- ETh Zurich, Zurich, Switzerland

REFERENCES:
- [Derived] Brnic M, Wegmuller R, Zeder C, Senti G, Hurrell RF. Influence of phytase, EDTA, and polyphenols on zinc absorption in adults from porridges fortified with zinc sulfate or zinc oxide. J Nutr. 2014 Sep;144(9):1467-73. doi: 10.3945/jn.113.185322. Epub 2014 Jun 25. PMID 24966411